CLINICAL TRIAL: NCT00696527
Title: National Prospective Survey on Women With a Diagnosis of Infiltrative Breast Cancer
Brief Title: National Survey on Infiltrative Breast Cancer
Acronym: CSI
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-OFR-DUM-2007/1
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Infiltrative Breast Cancer
Keywords: Infiltrative breast cancer-Clinical practice; Women with infiltrative breast cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this observational study is to describe radiological, clinical and histological characteristics of women with infiltrative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women> or = 18 years old
* Women with newly diagnosis of infiltrative breast cancer
* Agree to take part in this study

Exclusion Criteria:

* Women with other malignant tumor (except in situ cervical carcinoma or treated basal cell carcinoma)
* Women with in situ ductal carcinoma or in situ lobular carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First ten consecutive women with infiltrative breast cancer seen by oncologists, and fulfilling eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Radiological, Clinical and Histological characteristics | Once

SECONDARY OUTCOMES:
Treatments: Surgery, radiotherapy, chemotherapy, hormonotherapy. | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Medical Director, Study Director — AstraZeneca
Locations (107):
- France (107):
  - Research Site, Aix-en-Provence
  - Research Site, Alès
  - Research Site, Amilly
  - Research Site, Angers
  - Research Site, Annecy
  - Research Site, Arpajon
  - Research Site, Arras
  - Research Site, Aubervilliers
  - Research Site, Aulnay-sous-Bois
  - Research Site, Auxerre
  - Research Site, Avignon
  - Research Site, Beaune
  - Research Site, Besançon
  - Research Site, Béziers
  - Research Site, Bleriot
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Bruay-la-Buissière
  - Research Site, Bruges
  - Research Site, Caen
  - Research Site, Carcassonne
  - Research Site, Castelnau-le-Lez
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Chartre
  - Research Site, Cherbourg Octeville Cedex
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Colombes
  - Research Site, Coudekerque-Branche
  - Research Site, Créteil
  - Research Site, Croix
  - Research Site, Cucq
  - Research Site, Dax
  - Research Site, Dijon
  - Research Site, Évreux
  - Research Site, Grasse
  - Research Site, Grenoble
  - Research Site, Guilherand-Granges
  - Research Site, Hyères
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, La Garenne-Colombes
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Tronche
  - Research Site, Lagny-sur-Marne
  - Research Site, Le Chesnay
  - Research Site, Le Mans
  - Research Site, Lens
  - Research Site, Levallois-Perret
  - Research Site, Libourne
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Loos
  - Research Site, Lorient
  - Research Site, Lormont
  - Research Site, Lyon
  - Research Site, Mantes-la-Jolie
  - Research Site, Mareuil-lès-Meaux
  - Research Site, Marseille
  - Research Site, Meudon-la-Forêt
  - Research Site, Mont-de-Marsan
  - Research Site, Montmorency
  - Research Site, Montpellier
  - Research Site, Mulhouse
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Neuilly-sur-Seine
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Ploemeur
  - Research Site, Poissy
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Roanne
  - Research Site, Rodez
  - Research Site, Rouen
  - Research Site, Saint Mandee
  - Research Site, Saint-Benoît-la-Forêt
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Michel-sur-Orge
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saintes
  - Research Site, Sarcelles
  - Research Site, Sarcelle
  - Research Site, St.-Jean
  - Research Site, Strasbourg
  - Research Site, Thionville
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Troyes
  - Research Site, Valence
  - Research Site, Valenciennes
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vichy
  - Research Site, Villejuif